CLINICAL TRIAL: NCT06147882
Title: The Effect of Positive Psychotherapy-based Physicoeducation Program on Pain Perception , Activities of Daily Living, and Mental Health of Patients With Fibromyalgia Syndrome.
Brief Title: The Effect of Positive Psychotherapy Based Psychoeducation on Pain Perception With Fibromyalgia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Hamide Erol, PhD student, Duzce University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: duzceuniversityhamide001
Record Dates: First submitted 2023-10-06; First posted 2023-11-28 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Fibromyalgia Syndrome
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation Group (Active Comparator): The group of patients who are given psychoeducation program
  Interventions: Behavioral: The group will include patients with fibromyalgia syndrome who will receive positive psychotherapy.
- Control Group (No Intervention): The group of patients who are not given psychoeducation program

INTERVENTIONS:
Behavioral: The group will include patients with fibromyalgia syndrome who will receive positive psychotherapy. — The group will include patients with fibromyalgia syndrome who will receive positive psychotherapy.
  Arms: Psychoeducation Group

SUMMARY:
Fibromyalgia (FM) is characterized by symptoms such as chronic widespread pain, severe fatigue, sleep disturbances, extremity paresthesia, stiffness, mood disturbances, and cognitive impairment lasting more than 3 months without an alternative explanation. Although the exact etiology and pathogenesis of FM is still unknown, it has been suggested that stress or psychological factors may play a key role in the syndrome. 1,2,3 Positive Psychotherapy supports individuals in symptom management to use their resources to overcome difficulties, understand and recognize growth areas with a therapeutic approach.4 In this respect, it overlaps with the professional purpose of mental health and psychiatric nursing (RSPH). The aim of this study; In this study, it is aimed to report the process of examining the pain perception, daily life activities and mental health of patients with fibromyalgia syndrome (FMS) and the effectiveness of the psychoeducation program based on Positive Psychotherapy (PPT).

DETAILED DESCRIPTION:
The research is planned to be carried out between June 2023 and June 2024. The study will be conducted with patients diagnosed with FMS, who applied to a private Medical Center Orthopedics Outpatient Clinic in Düzce. The research was planned as a randomized controlled trial. The sample of the study will consist of patients selected by the randomization selection method who meet the inclusion criteria. The Gpower 3.1 program was used to determine the number of patients in the experimental and control groups of the study. In this context, two-way analysis of variance (TWO-WAY-ANOVA) method will be used. In conditions where the effect level was 0.40 (large effect), the error level (a) was 0.05, and the power of the test (1-B) was 0.95, the minimum sample size required for a statistically significant difference between the groups and between the measurements was obtained as 58. Each group must have at least 29 participants. In studies on the dependent variable in the literature, the drop out rate was found to be 6-12 (10-12%). Therefore, in this study, the drop out rate will be taken as 10, and the sample size will be determined as 34 for each group. The study was planned as 3 stages as randomized controlled pre-test, repeated post-test and 3rd month follow-up test. Within the scope of the study, Introductory Information Form, Visual Analogue Scale (VAS) (will be measured 3 times), Fibromyalgia Impact Questionnaire (FIQ) (will be measured 3 times), General Health Questionnaire-28 (GSA-28) (will be measured 3 times) will be applied. Within the scope of the research, it was planned to apply a PPT-based Psychoeducation Program consisting of 10 sessions, each of 120-90 minutes, to a group of participants diagnosed with FMS. The program to be implemented within the scope of the research was prepared after the literature review and together with the participant's handbook, it was sent to Positive Psychotherapy experts to get expert opinions. After the expert evaluations, necessary arrangements were made and the program was finalized. The applied Positive Psychotherapy group program was developed by the researcher by scanning the literature, the session contents, which blend three basic principles, including the real abilities of PPT, the balance model and the five-step therapy process, in order to minimize the symptoms that limit the daily life activities of FMS patients and create problems in their social lives. Information to be given, practices to be given and homework to be given for each session were determined. The purpose of the sessions was prepared by determining the targets expected to be achieved by the participants at the end of each session.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Having been diagnosed with Fibromyalgia Syndrome according to the 2016 ACR diagnostic criteria for at least 1 year,
* Agreeing to participate in the study.

Exclusion Criteria:

Those in acute depression

* History of a recent cardiac event such as myocardial infarction,
* History of significant head trauma,
* Peripheral neuropathy,
* Use of some centrally acting analgesic drugs such as opioids,
* History of substance and alcohol abuse,
* Concomitant autoimmune or inflammatory disease,
* Diseases affecting the central nervous system (for example, multiple sclerosis, Parkinson's disease),
* Serious psychiatric conditions that prevent participation (for example, psychotic disorders).
* Previously, therapy, counseling, personal development, etc. to have received

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Change in Pain Perception of Fibromyalgia Syndrome Patients from Baseline | Pre-test (Before positive psychotherapy group intervention), Post- test (10 weeks after therapy) and Follow up (12 weeks after therapy)
  Pain will be used to evaluate by VAS (Visual Anolog Scale) Line: A horizontal line is usually used, with the left end representing one extreme (e.g., "no pain" or "not at all") and the right end representing the other extreme (e.g., "worst pain imaginable" or "extremely intense").
  Length: The line is typically 100 millimeters long Participants are provided with instructions explaining what the scale measures (e.g., pain intensity) and are asked to mark a point on the line that best represents their experience.
  Scoring: Measurement is done by measuring the distance in millimeters from the left end of the line to the point marked by the participant. This provides a numerical score that quantifies the individual's perception.
  Interpretation: A higher score on the VAS generally indicates a more intense or severe experience of the measured phenomenon.
Change in daily living activities of fibromyalgia patients from baseline | Pre-test (Before positive psychotherapy group intervention), Post- test (10 weeks after therapy) and Follow up (12 weeks after therapy)
  Fibromyalgia Impact Questionnaire The Fibromyalgia Impact Questionnaire (FIQ) is a self-administered questionnaire designed to assess the health status and impact of fibromyalgia on individuals. It was developed to provide a comprehensive overview of the various aspects of fibromyalgia, including physical functioning, symptoms, and overall well-being.
  Physical Functioning:
  Work Status:
  Questions address how fibromyalgia affects an individual's ability to work.
  Depression and Anxiety:
  The FIQ includes questions about emotional well-being, assessing symptoms of depression and anxiety.
  Morning Tiredness:
  Measures the level of fatigue and tiredness experienced in the morning, providing insights into the impact of fibromyalgia on sleep and morning functioning.
  Pain Levels:
  Questions related to the intensity of pain experienced by individuals with fibromyalgia.
  Stiffness:
  Assesses the extent of stiffness experienced by individuals, which is a common symptom of fibromyalgia.

SECONDARY OUTCOMES:
Change in the mental health of fibromyalgia patients from the beginning | Pre-test (Before positive psychotherapy group intervention), Post- test (10 weeks after therapy) and Follow up (12 weeks after therapy)
  General Health Questionnaire-28 General Health Questionnaire -28 is a self-filled screening test designed to detect mental health problems encountered in society and non-psychiatric clinical settings. The survey consists of four subsections, each consisting of seven items. These sections; Somatic symptoms include anxiety and sleep disorders, impairment in social functioning, and major depression. The 28-item scale consists of a question about whether each individual has a recent complaint and a four-item response ranging from "less than usual" to "much more than usual". After the application, a minimum score of 0 and a maximum of 28 points can be obtained, and a higher score increases the likelihood of mental health disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Düzce Üniversitesi, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erol H, Karaca A. The Effect of Positive Psychotherapy on Pain Perception, Daily Functioning, and Mental Health in Patients With Fibromyalgia. Pain Manag Nurs. 2025 Dec;26(6):e550-e560. doi: 10.1016/j.pmn.2025.07.007. Epub 2025 Sep 4. PMID 40912975